CLINICAL TRIAL: NCT02156492
Title: A Pharmacokinetic, Pharmacodynamic, and Drug-Drug Interaction Study of Evacetrapib With Selected Statins in Healthy Chinese Subjects
Brief Title: A Study of Evacetrapib With Selected Statins in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14467; I1V-MC-EIAM (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-28; First posted 2014-06-05 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Simvastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Evacetrapib Single (Experimental): Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
  Interventions: Drug: Evacetrapib
- Evacetrapib Multiple (Experimental): Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib for 14 days.
  Interventions: Drug: Evacetrapib
- Simvastatin (Active Comparator): Part 2, Cohorts B, Participants will receive simvastatin orally, once daily on Days 1 - 4.
  Interventions: Drug: Simvastatin
- Evacetrapib and Simvastatin (Experimental): Part 2, Cohorts B, Participants will receive evacetrapib orally once daily on Days 5 - 14 and simvastatin orally, once daily on Days 15 - 22.
  Interventions: Drug: Evacetrapib; Drug: Simvastatin
- Atorvastatin (Active Comparator): Part 2, Cohorts C, Participants will receive atorvastatin orally, once daily on Days 1 - 4.
  Interventions: Drug: Atorvastatin
- Evacetrapib and Atorvastatin (Experimental): Part 2, Cohorts C, Participants will receive evacetrapib orally once daily on Days 5 - 14 and atorvastatin orally, once daily on Days 15 - 22.
  Interventions: Drug: Evacetrapib; Drug: Atorvastatin

INTERVENTIONS:
Drug: Evacetrapib — Administered orally.
  Other Names: LY2484595
  Arms: Evacetrapib Multiple; Evacetrapib Single; Evacetrapib and Atorvastatin; Evacetrapib and Simvastatin
Drug: Simvastatin — Administered orally.
  Arms: Evacetrapib and Simvastatin; Simvastatin
Drug: Atorvastatin — Administered orally.
  Arms: Atorvastatin; Evacetrapib and Atorvastatin

SUMMARY:
The main purpose of this study is to investigate how the body responds to evacetrapib and to evaluate the safety and the effect of evacetrapib, alone and in combination with selected statins, in healthy Chinese participants. The study has 2 parts. Part one will last up to 4 weeks and part two will last up to 5 weeks, not including screening. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese and living in China.
* Are overtly healthy males or females as determined by medical history and physical examination.
* Female participants:

  * Women not of child-bearing potential
  * Women of child-bearing potential must correctly use 2 forms of reliable contraception to avoid getting pregnant during the study and for 3 months after the study is completed.
* Body Mass Index: 19.0 to 24.0 kilogram per square meter (kg/m^2)
* BP and pulse rate at both supine and standing positions of approximately a systolic BP ≤ 140 millimeter of mercury (mm Hg), and diastolic BP ≤ 90 mm Hg
* Participants with untreated hypercholesterolemia may be included if not on an herbal or other traditional Chinese medicines (TCM)
* Have no known liver disease
* Have given written informed consent

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product (IP) or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to evacetrapib, simvastatin, or atorvastatin, related compounds or any components of the formulation
* Have previously completed or withdrawn from this study or any other study investigating evacetrapib, and have previously received the IP within 3 months.
* Have a history within the last year or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurologic disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Show evidence of significant active neuropsychiatric disease.
* Regularly use known drugs of abuse
* Are women with a positive pregnancy test or women who are lactating.
* Have used or intend to use over-the-counter or prescription medications (including vitamins/mineral supplements) or TCM 14 days prior to the first dose and during the study.

  * Hormonal contraceptives are permitted.
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of organic anion transporting polypeptide 1B1 (OATP1B1), or of any other transporters involved in simvastatin or atorvastatin disposition, or of any drugs or substances that are known to be strong inducers or inhibitors of cytochrome P450 3A (CYP3A) within 30 days prior to the first dose and throughout the study.
* Donated blood of >400 mL within the last month.
* Drink alcoholic beverages with intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption 48 hours prior to dosing until discharge from the clinical research unit (CRU) (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Are unwilling to comply with the dietary requirements/restrictions during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Evacetrapib Single and Multiple Dose: Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
  Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib 130 mg for 14 days.
- Cohort B: Evacetrapib and Simvastatin: Part 2, Cohorts B, Period 1, Participants will receive simvastatin 40 mg orally, once daily on Days 1 - 4
  Part 2, Cohorts B, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohorts B, Period 3, Participants will receive evacetrapib 130 mg and simvastatin 40mg orally, once daily on Days 15 - 22.
- Cohort C: Evacetrapib and Atorvastatin: Part 2, Cohorts C, Period 1, Participants will receive atorvastatin orally, once daily on Days 1 - 4.
  Part 2, Cohorts C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohorts C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
Period: Period 1
Arm/Group | Cohort A: Evacetrapib Single and Multiple Dose | Cohort B: Evacetrapib and Simvastatin | Cohort C: Evacetrapib and Atorvastatin
Started | 16 | 24 | 22
Received at Least One Dose of Study Drug | 16 | 24 | 22
Completed | 16 | 23 | 22
Not Completed | 0 | 1 | 0
Not completed — No Reason Given | 0 | 1 | 0
Period: Period 2
Arm/Group | Cohort A: Evacetrapib Single and Multiple Dose | Cohort B: Evacetrapib and Simvastatin | Cohort C: Evacetrapib and Atorvastatin
Started | 16 | 23 | 22
Completed | 16 | 23 | 22
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort A: Evacetrapib Single and Multiple Dose | Cohort B: Evacetrapib and Simvastatin | Cohort C: Evacetrapib and Atorvastatin
Started | 0 (Cohort A participated in Period 1 and Period 2 only.) | 23 | 22
Completed | 0 | 22 | 22
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Cohort A: Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
  Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib 130 mg for 14 days.
- Cohort B: Part 2, Cohorts B, Period 1, Participants will receive simvastatin 40 mg orally, once daily on Days 1 - 4.
  Part 2, Cohorts B, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohorts B, Period 3, Participants will receive evacetrapib 130 mg and simvastatin 40mg orally, once daily on Days 15 - 22.
- Cohort C: Part 2, Cohorts C, Period 1, Participants will receive atorvastatin orally, once daily on Days 1 - 4.
  Part 2, Cohorts C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohorts C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 16 | 24 | 22 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (8.0) | 27.5 (2.9) | 27.9 (4.9) | 28.02 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 5
  Male | 13 | 24 | 20 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 16 | 24 | 22 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 16 | 24 | 22 | 62

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under Curve (AUC 0-inf) of Evacetrapib
Description: Pharmacokinetic (PK) parameter estimates from evacetrapib concentrations following single dose and daily dose of 130 mg evacetrapib.
Time Frame: Part 1: Day 1 Predose 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144, and 168 hours Postdose; Part 2 Day 14 Predose 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours Postdose
Population: All participants who received at least one dose of study drug in Cohort A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Groups:
- Evacetrapib Single and Multiple Dose: Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
  Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib 130 mg for 14 days.
Arm/Group | Evacetrapib Single and Multiple Dose
Number analyzed (Participants) | 16
nanogram * hour per milliliter (ng*h/mL)
  Day 1 | 7700 (74)
  Day 14 | 23600 (33)

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Evacetrapib
Description: Pharmacokinetic parameter estimates from evacetrapib following single dose and daily doses of 130 mg.
Time Frame: Part 1: Day 1 and Day 14 Predose 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144, and 168 hours Postdose; Part 2 Day 14: Predose 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours Postdose
Population: All participants who received at least one dose of study drug in Cohort A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Evacetrapib Single and Multiple Dose
Number analyzed (Participants) | 16
ng/mL
  Single Dose Day 1 | 418 (118)
  Multiple Dose Day 14 | 954 (52)

3. Primary Outcome: PK: Time to Maximum Concentration (Tmax) of Evacetrapib
Description: Pharmacokinetic parameter estimates of evacetrapib following single and daily doses of 130 mg evacetrapib.
Time Frame: Part 1: Day 1 Predose on Day 1 or Day 14 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144, and 168 hours postdose. Part 2: Predose on Day 14 at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours post dose.
Population: All participants who received at least one dose of study drug in Cohort A.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Evacetrapib Single and Multiple Dose
Number analyzed (Participants) | 16
hours (h)
  Single Dose Day 1 | 3.00 [2.00 to 6.00]
  Daily Dose Day 14 | 3.00 [2.00 to 4.00]

4. Primary Outcome: PK: AUC of Evacetrapib Alone and With Simvastatin or Atorvastatin
Description: Pharmacokinetic parameter estimates of evacetrapib following 130 mg evacetrapib daily alone or with 40 mg simvastatin or 20 mg atorvastatin daily AUC (0-24).
Time Frame: Part 2: Day 14 and 22 Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours Postdose
Population: All participants who received at least one dose of study drug in Cohort B and C and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Evacetrapib Daily and Simvastatin: Part 2, Cohorts B, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14.
  Part 2, Cohorts B, Period 3, Participants will receive evacetrapib 130 mg and simvastatin 40mg orally, once daily on Days 15 - 22.
- Evacetrapib Daily and Atorvastatin: Part 2, Cohorts C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14.
  Part 2, Cohorts C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
Arm/Group | Evacetrapib Daily and Simvastatin | Evacetrapib Daily and Atorvastatin
Number analyzed (Participants) | 23 | 22
ng*h/mL
  Days 5-14 | 10700 (36) | 10600 (30)
  Days 15-22 | 9640 (48) | 9480 (53)

5. Primary Outcome: PK: Cmax of Evacetrapib Alone and With Simvastatin or Atorvastatin
Description: Pharmacokinetic parameter estimates of evacetrapib following 130 mg evacetrapib daily alone or with 40 mg simvastatin or 20 mg atorvastatin daily.
Time Frame: Part 2: Day 14 and 22 Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours Postdose.
Population: All participants who received at least one dose of study drug in Cohort B and C and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Evactrapib Daily and Atorvastatin: Part 2, Cohorts C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14.
  Part 2, Cohorts C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
Arm/Group | Evacetrapib Daily and Simvastatin | Evactrapib Daily and Atorvastatin
Number analyzed (Participants) | 23 | 22
ng/mL
  Days 5-14 | 1180 (52) | 1120 (36)
  Days 15- 22 | 1020 (68) | 1000 (73)

6. Primary Outcome: PK: Tmax of Evacetrapib Alone and With Simvastatin or Atorvastatin
Description: Pharmacokinetic parameter estimates of Tmax of evacetrapib following 130 mg daily dose alone or with 40 mg Simvastatin or 20 mg Atorvastatin. Tmax of simvastatin and atorvastatin.
Time Frame: Part 2: Predose on Day 14 and 22 and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours postdose.
Population: All participants who received at least one dose of study drug in Cohort B and C and had evaluable PK data.
Measure: Median (Full Range); unit: h
Groups:
- Evacetrapib Daily and Simvastatin: Part 2, Cohorts B, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohorts B, Period 3, Participants will receive evacetrapib 130 mg and simvastatin 40mg orally, once daily on Days 15 - 22.
- Evacetrapib Daily and Atrovastatin: Part 2, Cohort C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
  Part 2, Cohort C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
Arm/Group | Evacetrapib Daily and Simvastatin | Evacetrapib Daily and Atrovastatin
Number analyzed (Participants) | 23 | 22
h
  Days 5-14 | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 6.00]
  Days 15- 22 | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00]

7. Secondary Outcome: Effect of Evacetrapib Single and Multiple Doses on High Density Lipoprotein Cholesterol (HDL-C), Low Density Lipoprotein Cholesterol (LDL-C), and Triglycerides (TG)
Time Frame: Single Dose Day 2 and Multiple Dose Day 22
Population: All participants who received at least one dose of study drug in Cohort A.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Groups:
- Evacetrapib Single Dose Day 2: Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
- Evacetrapib Multiple Dose Day 22: Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib 130 mg for 14 days.
Arm/Group | Evacetrapib Single Dose Day 2 | Evacetrapib Multiple Dose Day 22
Number analyzed (Participants) | 16 | 16
millimoles per liter (mmol/L)
  HDL-C | 1.641 (0.211) | 2.676 (0.373)
  LDL-C | 2.289 (0.483) | 1.241 (0.574)
  TG | 0.984 (0.312) | 1.221 (0.356)

ADVERSE EVENTS:
Groups:
- Evacetrapib Single Cohort A: Part 1, Cohort A, Period 1, Participants will receive a single oral 130 mg dose of evacetrapib.
- Evacetrapib Multiple: Part 1, Cohort A, Period 2, Participants will receive multiple doses of evacetrapib 130 mg for 14 days.
- Simvastatin: Part 2, Cohorts B, Period 1, Participants will receive simvastatin 40 mg orally, once daily on Days 1 - 4.
- Evacetrapib Single Cohort B: Part 2, Cohorts B, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
- Evacetrapib and Simvastatin: Part 2, Cohorts B, Period 3, Participants will receive evacetrapib 130 mg and simvastatin 40mg orally, once daily on Days 15 - 22.
- Atorvastatin: Part 2, Cohorts C, Period 1, Participants will receive atorvastatin orally, once daily on Days 1 - 4.
- Evacetrapib Single Cohort C: Part 2, Cohorts C, Period 2, Participants will receive a single oral 130 mg dose of evacetrapib on Days 5-14
- Evacetrapib and Atorvastatin: Part 2, Cohorts C, Period 3, Participants will receive evacetrapib 130 mg orally and atorvastatin 20 mg orally, once daily on Days 15 - 22.
Arm/Group | Evacetrapib Single Cohort A | Evacetrapib Multiple | Simvastatin | Evacetrapib Single Cohort B | Evacetrapib and Simvastatin | Atorvastatin | Evacetrapib Single Cohort C | Evacetrapib and Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/24 | 0/23 | 0/23 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/24 | 0/23 | 0/23 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No